CLINICAL TRIAL: NCT04934150
Title: Neuronavigated Repetitive Transcranial Magnetic Stimulation (nrTMS) of the Dorsolateral Prefrontal and Primary Motor Cor-tex for the Treatment of Chronic Pain: a Randomized Place-bo-controlled Trial
Brief Title: Neuronavigated Repetitive Transcranial Magnetic Stimulation (nrTMS) of the Dorsolateral Prefrontal and Primary Motor Cortex for the Treatment of Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 30-459-ex 17/18
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: The study was conducted in a single-blinded, randomized, placebo-controlled design
Who Masked: Participant
Masking Description: Sham stimulation was provided by turning the TMS coil to the non-stimulating side.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- M1 stimulation (Active Comparator): 10 Hz stimulation of left motor area
  Interventions: Device: navigated repetitive Transcranial Stimulation
- DLPFC stimulation (Active Comparator): 5 Hz stimulation of left dorsolateral prefrontal cortex
  Interventions: Device: navigated repetitive Transcranial Stimulation
- Sham TMS (Sham Comparator): Sham TMS over the left M1 area
  Interventions: Device: navigated repetitive Transcranial Stimulation

INTERVENTIONS:
Device: navigated repetitive Transcranial Stimulation — High frequency nrTMS over 13 sessions (1800-2000 pulses per session) over DLPFC and M1 cortical areas.

SUMMARY:
This study investigated the effects of navigated repetitive Transcranial Magnetic Stimulation on nociception and quality of life in patients suffering from chronic pain conditions. Two cortical targets (dorsolateral prefrontal cortex/DLPFC and M1 area) were stimulated and compared to Sham stimulation.

DETAILED DESCRIPTION:
From 34 patients, 24 completed the study. The M1-area was stimulated with 10 Hz rTMS while the DLPFC received a 5Hz stimulation. In total, 13 session were administered over a period of 36 weeks with most frequent stimulation in the first 4 weeks of the trial. Results were compared to Sham-TMS over the M1 area at the same schedule than the actual therapy. Outcome parameters included the German Pain Questionnaire (GPQ), the Depression, Anxiety and Stress Scale" (DASS) and quality of life (QoL) with the SF-12 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years
* clinical diagnosis of chronic LBP (low back pain) and or neck pain
* average resting pain-level > than 3 in the Numeric Rating Scale (0-10)
* no changes in pain medication 4 weeks at baseline
* no surgical procedures in the last 2 years

Exclusion Criteria:

* metallic and electronic implants in the head, neck and chest
* medication e.g. tetracyclic antidepressants, antiviral, antipsychotic, opioid doses > 100mg orally/d
* history of frequent headache or tinnitus
* alcohol or drug abuse
* pregnant patients
* breastfeeding patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale | 36 weeks
  0-10 0 = no pain, 10 = worst pain

SECONDARY OUTCOMES:
Self-reported "Depression, Anxiety and Stress Scale" (DASS) questionnaire. | 36 weeks
  0- 21 for each item, higher scores indicate worse symptoms. Lower scores indicate a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No